CLINICAL TRIAL: NCT07130110
Title: Diagnostic Contribution of Bronchoalveolar Lavage to Lung Cryotransbronchial Biopsy in Interstitial Lung Diseases
Brief Title: BAL Contribution to Lung Cryo-TBB in ILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Yedikule Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ERDOGAN CETINKAYA, Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cryobiopsy+BAL
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Bronchoalveolar Lavage (BAL); Transbronchial Cryobiopsy; Interstitial Lung Disease (ILD)
Keywords: Interstitial Lung Disease; Bronchoalveolar lavage; Cryotransbronchial biopsy
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research group (Experimental): A group investigating the contribution of bronchoalveolar lavage to the diagnosis in patients undergoing cryo-transbronchial biopsy for interstitial lung diseases
  Interventions: Diagnostic Test: Transbronchial cryobiopsy; Diagnostic Test: Bronchoalveolar Lavage

INTERVENTIONS:
Diagnostic Test: Transbronchial cryobiopsy — The c-TBB procedure was performed under general anesthesia with rigid bronchoscopy guidance. The biopsy site was selected based on the area of highest involvement seen on thoracic CT. After evaluating the trachea and main bronchi with a rigid bronchoscope, a flexible bronchoscope was advanced into the target segment. Using a 1.9 mm, 90 cm cryoprobe, tissue was frozen and rapidly retracted with the bronchoscope to obtain the biopsy. The specimen was placed in formalin without damage. Hemorrhage control was achieved with a Fogarty balloon. A chest X-ray was taken two hours later to check for pneumothorax risk.
Diagnostic Test: Bronchoalveolar Lavage — The BAL protocol, including pre-procedural preparations and the procedure itself, was performed in accordance with the American Thoracic Society (ATS) guidelines. In cases of diffuse involvement, BAL was performed from the middle lobe or lingula, while in localized involvement, it was done from the affected area. The target segment was occluded with the bronchoscope, and room-temperature 0.9% NaCl solution was instilled in 20 cc portions and gently aspirated to prevent airway collapse. A minimum of 100 mL (maximum 300 mL) saline was used, with at least 30% recovery required. Cellular analysis of BAL fluid was conducted per ATS guidelines. Normal cell distribution: alveolar macrophages >85%, lymphocytes 10-15%, neutrophils ≤3%, eosinophils ≤1%, squamous/ciliated columnar epithelial cells ≤1%.

SUMMARY:
The goal of this observational study is to evaluate whether performing bronchoalveolar lavage (BAL) simultaneously with transbronchial lung cryobiopsy (c-TBB) can improve diagnostic yield in adult patients with suspected interstitial lung disease (ILD).

The main questions it aims to answer are:

* Does the addition of BAL to c-TBB increase the overall diagnostic accuracy in ILD patients?
* Can the combination of BAL and c-TBB reduce the need for surgical lung biopsy in the diagnostic process of ILD?

If there is a comparison group: Researchers will compare patients diagnosed by c-TBB alone to those evaluated with both c-TBB and BAL to see if BAL provides additional diagnostic value, especially in cases where histopathological findings from c-TBB are inconclusive.

Participants will:

Undergo transbronchial lung cryobiopsy (c-TBB) under general anesthesia to collect lung tissue samples.

Have bronchoalveolar lavage (BAL) performed in the same session using ATS guideline-based protocols.

Be evaluated in a multidisciplinary discussion (MDD) integrating clinical, radiologic, and pathologic findings to establish a final diagnosis.

DETAILED DESCRIPTION:
Interstitial Lung Diseases (ILDs) are a rare group of diseases characterized by inflammation and fibrosis of the lung interstitium, with many subtypes. The incidence is reported as approximately 75 per 100,000 in the US and Europe, and 25.8 in Turkey. ILDs are classified into known causes, idiopathic interstitial pneumonias (IIPs), granulomatous diseases, and other subgroups.

While surgical lung biopsy remains the gold standard for diagnosis, it carries risk of complications. Therefore, cryobiopsy (c-TBB), a minimally invasive method, is preferred, with diagnostic yield ranging between 50-90%.

Bronchoalveolar lavage (BAL) provides cellular analysis from the alveoli, aiding differential diagnosis in ILD but is limited as a sole diagnostic tool. Combined use of c-TBB and BAL may improve diagnostic accuracy and reduce the need for surgical biopsy.

In this study, the diagnostic contribution of simultaneous BAL in patients undergoing c-TBB with a preliminary ILD diagnosis was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 18,
* Patients diagnosed with interstitial lung disease through imaging methods, and patients who underwent cryotransbronchial biopsy and bronchoalveolar lavage

Exclusion Criteria:

* Being under 18 years of age,
* Patients diagnosed with malignancy,
* Patients who underwent non-standardized bronchoalveolar lavage,
* Patients whose data are unavailable

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield of c-TBB | Within 1 week after the procedure
  The proportion of patients in whom a histopathological diagnosis was established using transbronchial cryobiopsy (c-TBB).

SECONDARY OUTCOMES:
Contribution of BAL to Multidisciplinary Diagnosis (MDD) | Within 1 month of the procedure
  The proportion of cases where bronchoalveolar lavage (BAL) provided additional diagnostic value in reaching a final diagnosis during multidisciplinary discussion.
Diagnostic Yield of Multidisciplinary Discussion in c-TBB-Negative Cases | Within 1 month of the procedure
  The number and percentage of patients without histopathological diagnosis via c-TBB who were subsequently diagnosed through MDD.
Procedure-Related Complications of c-TB | Within 48 hours after the procedure
  The rate and type of complications observed following the c-TBB procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Kazlıçeşme Mh, Belgrad Kapı yolu Cad No:1, 34020 Zeytinburnu/İstanbul, Istanbul, Turkey (Türkiye)